CLINICAL TRIAL: NCT02586454
Title: Transmuscular Quadratus Lumborum Block for Postoperative Pain After Total Abdominal Hysterectomy
Brief Title: Analgesic Efficacy of Transmuscular Quadratus Lumborum in Patients Undergoing Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuala Lumpur General Hospital (Other Government)
Responsible Party: Principal Investigator, Amiruddin Nik Mohamed Kamil, Dr, Kuala Lumpur General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-15-919-25992
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Pain Postoperative
Keywords: Transmuscular quadratus lumborum block, total abdominal hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transmuscular quadratus lumborum (QL) block (Experimental): Bilateral QL block using 20 ml 0.375% ropivacaine in each side (to a maximum dose 3 mg/kg) plus patient controlled analgesia morphine (1mg/bolus morphine, lockout time 5 minutes) post operative
  Interventions: Procedure: Transmuscular quadratus lumborum block; Drug: morphine; Drug: ropivacaine
- Control (Active Comparator): Patient controlled analgesia morphine (1mg/bolus morphine, lockout time 5 minutes) post operative
  Interventions: Drug: morphine

INTERVENTIONS:
Procedure: Transmuscular quadratus lumborum block
  Arms: Transmuscular quadratus lumborum (QL) block
Drug: morphine
Drug: ropivacaine
  Arms: Transmuscular quadratus lumborum (QL) block

SUMMARY:
Patients who have undergone laparotomies often require multimodal postoperative pain regimes. In recent years, abdominal wall blocks have been included to become part of this in order to overcome side effects of systemic opioids and complications from epidural analgesia.

Borglum popularised a new approach on abdominal wall blocks by introducing the transmuscular quadratus lumborum (QL) block. Transmuscular QL block is thought to be effective against somatic and visceral pain as local anaesthetic tends to spread from the site of injection to thoracic paravertebral spaces where the sympathetic chain lies.

The objective of this study is to evaluate the analgesic efficacy of transmuscular QL block in patients undergoing total abdominal hysterectomy (TAH) by measuring cumulative opioid consumption, pain score at rest and on movement 24 hours after TAH. Our hypothesis is patients given transmuscular QL block will have lower cumulative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II
2. Patient's weight > 50kg
3. Elective TAH

Exclusion Criteria:

1. Body mass index (BMI) > 35 kg/m2
2. Any contraindications to peripheral nerve blocks i.e. local skin infection, coagulopathy, allergy to LA
3. Inability to use patient controlled analgesia
4. Patient on antiplatelet, anticoagulant or on regular use of opioids, paracetamol, nonsteroidal anti-inflammatory drugs or tramadol for chronic condition

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption | 24 hours after total abdominal hysterectomy
  in mg for 24 hours
Pain score at rest and movement | 24 hours after total abdominal hysterectomy
  using visual analogue scale 1 to 10

SECONDARY OUTCOMES:
Complications related to the transmuscular QL block | 24 hours after total abdominal hysterectomy
  Complications related to transmuscular QL block: Haematoma at site of injection,infection at site of injection Complications related to PCAM:Nausea, vomiting, pruritus, sedation

CONTACTS AND LOCATIONS:
Overall Officials: Amiruddin Nik Mohamed Kamil, MBBS MMed (Anaesthesiology), Principal Investigator — Kuala Lumpur General Hospital
Locations (1):
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Kadam VR. Ultrasound guided quadratus lumborum block or posterior transversus abdominis plane block catheter infusion as a postoperative analgesic technique for abdominal surgery. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):130-1. doi: 10.4103/0970-9185.150575. No abstract available. PMID 25788791
- [Background] Visoiu M, Yakovleva N. Continuous postoperative analgesia via quadratus lumborum block - an alternative to transversus abdominis plane block. Paediatr Anaesth. 2013 Oct;23(10):959-61. doi: 10.1111/pan.12240. Epub 2013 Aug 9. PMID 23927552
- See also: Related Info — http://cdn.intechopen.com/pdfs/38231/InTech-Abdominal_surgery_advances_in_the_use_of_ultrasound_guided_truncal_blocks_for_perioperative_pain_management.pdf